CLINICAL TRIAL: NCT00267813
Title: The Effects of Craving and Abstinence From Cigarettes on Brain Metabolism in Smokers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Aviv M. Weinstein, Sourasky Medical Center Tel Aviv
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-O5-EE-065-CTIL
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Nicotine Dependence
Keywords: craving; nicotine; imaging; FDG; PET; smoking; Bupropion
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bupropion (Zyban) — 1 tablet a day increasing to 2 tablets a day after a week

SUMMARY:
Craving and withdrawal from smoking cigarettes are major factors for relapse. We investigated craving for cigarettes in smokers undergoing pharmacological treatment with Bupropion (Zyban). We compare cue-induced reactivity to smoking videos in smokers who were successfully treated with Bupropion to smokers who are still smoking. We measured the brain's metabolic activity in response to smoking and neutral cues in Positron Emission Tomography using FDG.

DETAILED DESCRIPTION:
Craving and withdrawal from smoking cigarettes are major factors for relapse. We investigated craving for cigarettes in smokers undergoing pharmacological treatment with Bupropion (Zyban)for 2 months. We compare cue-induced reactivity to smoking videos in smokers who were successfully treated with Bupropion to smokers who are still smoking. We measured the brain's metabolic activity after exposure to videotapes showing smoking and neutral scenes in Positron Emission Tomography using FDG. There were 2 scanning sessions, one with a smoking videotape and one with a neutral video separated by a week. So far we have compared the brain's metabolic activity in 6 abstinent smokers and 6 still smokers.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smokers (over 1 pack a day)
* Age 20-65, male-females

Exclusion Criteria:

* Dependence on other substances
* Psychiatric diagnosis
* Neurological disorder
* Obesity
* Young persons
* Pregnant women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Brain metabolic activity (FDG) in response to craving and neutral cues. | 30-40 minutes

SECONDARY OUTCOMES:
Subjective ratings of craving | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even-Sapir, M.D, Ph.D, Principal Investigator — Tel-Aviv Sourasky Medical Center; Aviv M Weinstein, Ph.D, Principal Investigator — Tel-Aviv Sourasky Medical Center; Hedva Lerman, M.D, Study Director — Tel-Aviv Sourasky Medical Center
Locations (1):
- Department of Nuclear Medicine, Tel Aviv, Israel

REFERENCES:
- [Derived] Weinstein A, Greif J, Yemini Z, Lerman H, Weizman A, Even-Sapir E. Attenuation of cue-induced smoking urges and brain reward activity in smokers treated successfully with bupropion. J Psychopharmacol. 2010 Jun;24(6):829-38. doi: 10.1177/0269881109105456. Epub 2009 Jul 31. PMID 19648219